CLINICAL TRIAL: NCT05886569
Title: Edge AI-deployed DIGItal Twins for PREDICTing Disease Progression and Need for Early Intervention in Infectious and Cardiovascular Diseases Beyond COVID-19 - Evaluation of Physiological Sensors
Brief Title: DIGIPREDICT-Physio-DE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Laurenz Kopp Fernandes, Senior physician, Transplant Outpatient Unit, Charite University, Berlin, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DIGIPREDICT-Physio-DE
Record Dates: First submitted 2023-05-12; First posted 2023-06-02 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Biomarkers
Keywords: Bioimpedance; Body surface temperature; Blood count; C-reactive protein; Ferritin; high sensitive Troponin T; Interleukin-6; Lactate; NT-proBNP; pH; Procalcitonin; Kinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional group (Experimental): This arm includes all study participants.
  Interventions: Device: DIGIPREDICT Physiopatech

INTERVENTIONS:
Device: DIGIPREDICT Physiopatech — Application of the DIGIPREDICT Physiopatch investigational device

SUMMARY:
The study aims to investigate short-term physiological and biochemical inflammatory and cardiocirculatory biomarker kinetics in heart failure patients, using the DIGIPREDICT Physiopatch device - an investigational device that allows non-invasive realtime single-lead ECG registration and bioimpedance measurement as well as spotcheck photoplethysmography -, and standard laboratory methods, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Presence of heart failure, defined as: symptoms and signs of heart failure, elevated baseline NT-proBNP levels (>125pg/ml in sinus rhythm, >365 pg/ml in atrial fibrillation) without severe kidney disease (defined as eGFR(MDRD)<30 ml/min/1.73m²), and structural and/or functional abnormalities (according to 2021 ESC Heart Failure Guidelines)
* At least 2 days of further treatment on a DHZC intensive care unit (H3i, IPS1, IPS2) or intermediate care unit (H3 - heart failure unit) expected at enrolment.
* Age of subject is ≥ 18years.
* Subject is female, male, divers.
* Signed written informed consent.
* For female subject or divers subject:

  1. Negative highly sensitive urine or serum pregnancy test before inclusion, and
  2. Practicing a highly effective birth control method (failure rate of less than 1%):

     1. combined (estrogen and progestogen containing) hormonal
     2. contraception associated with inhibition of ovulation (oral/intravaginal/ transdermal), or
     3. progestogen-only hormonal contraception associated with inhibition of ovulation (oral/injectable/implantable), or
     4. intrauterine device (IUD), or
     5. intrauterine hormone-releasing system ( IUS), or
     6. bilateral tubal occlusion, or
     7. vasectomised partner, or
     8. heterosexual abstinence.

Exclusion Criteria:

* Subject is breastfeeding.
* Subject suffers from an addiction or from a disease that prevents the subject from recognizing nature, scope, and consequences of the study.
* Subject is treated with immunosuppressive drugs at enrolment.
* Subject requires mechanical circulatory support at enrolment (IABP, veno-arterial ECMO, Impella, VAD, TAH).
* Subject requires extracorporeal lung support at enrolment (veno-venous ECMO, interventional lung assist).
* Subject requires invasive ventilation at enrolment.
* Subject requires renal replacement therapy.
* Subjects with an active stimulation device (implanted or not) (e.g. pacemaker, nerve stimulator).
* Subject has a known colonisation or infection with multi-drug-resistant pathogens.
* Subject suffers from a skin disease at all possible placement sites for the DIGIPREDICT Physiopatch.

Subject has damaged skin at all fingertips.

* Subject has highly sensitive skin to (medical) adhesives.
* Subject shows an inability to comply with all of the study procedures and follow-up visits.
* Subjects who are unwilling to consent to saving and propagation of pseudonymised medical data for study reasons.
* Subject is legally detained in an official institution.
* Subject is dependent on the sponsor, the investigator or the study sites.
* Subject participates in another clinical investigation according to MPDG/MDR, or in a study according to AMG/CTR that investigates immunosuppressive drugs at the time of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-05-25 (Estimated); Primary Completion 2023-11-24 (Estimated); Study Completion 2023-11-24 (Estimated)

PRIMARY OUTCOMES:
Short-term kinetics of C-reactive protein | 4 days
  Outcome is the detection of kinetics of C-reactive protein values [mg/L] between at least two timestamps.
  Short-term is defined as <= 26hours; biomarker kinetics are defined as >20% increase or decrease of a biomarker level at one point in time compared to the level at another point in time. The timestamp documented in the electronic health record will be used for analysis.
Short-term kinetics of procalcitonin | 4 days
  Outcome is the detection of kinetics of procalcitonin values [ng/mL] between at least two timestamps.
  Short-term is defined as <= 26hours; biomarker kinetics are defined as >20% increase or decrease of a biomarker level at one point in time compared to the level at another point in time. The timestamp documented in the electronic health record will be used for analysis.
Short-term kinetics of interleukin-6 | 4 days
  Outcome is the detection of kinetics of interleukin-6 values [ng/L] between at least two timestamps.
  Short-term is defined as <= 26hours; biomarker kinetics are defined as >20% increase or decrease of a biomarker level at one point in time compared to the level at another point in time. The timestamp documented in the electronic health record will be used for analysis.
Short-term kinetics of ferritin | 4 days
  Outcome is the detection of kinetics of ferritin values [µg/L] between at least two timestamps.
  Short-term is defined as <= 26hours; biomarker kinetics are defined as >20% increase or decrease of a biomarker level at one point in time compared to the level at another point in time. The timestamp documented in the electronic health record will be used for analysis.
Short-term kinetics of NT-pro brain natriuretic peptide | 4 days
  Outcome is the detection of kinetics of NT-pro brain natriuretic peptide [ng/L] between at least two timestamps.
  Short-term is defined as <= 26hours; biomarker kinetics are defined as >20% increase or decrease of a biomarker level at one point in time compared to the level at another point in time. The timestamp documented in the electronic health record will be used for analysis.
Short-term kinetics of high sensitive troponin T | 4 days
  Outcome is the detection of kinetics of high sensitive troponin T [ng/L] between at least two timestamps.
  Short-term is defined as <= 26hours; biomarker kinetics are defined as >20% increase or decrease of a biomarker level at one point in time compared to the level at another point in time. The timestamp documented in the electronic health record will be used for analysis.
Short-term kinetics of lactate | 4 days
  Outcome is the detection of kinetics of lactate [mg/dL] between at least two timestamps.
  Short-term is defined as <= 26hours; biomarker kinetics are defined as >20% increase or decrease of a biomarker level at one point in time compared to the level at another point in time. The timestamp documented in the electronic health record will be used for analysis.
Short-term kinetics of blood pH | 4 days
  Outcome is the detection of kinetics of blood pH between at least two timestamps.
  Short-term is defined as <= 26hours; biomarker kinetics are defined as >20% increase or decrease of a biomarker level at one point in time compared to the level at another point in time. The timestamp documented in the electronic health record will be used for analysis.
Short-term kinetics of body surface temperature | 4 days
  Outcome is the detection of kinetics of body surface temperature [°C] between at least two timestamps. The mean value within 1 h before the timestamp of the concomitant biochemical biomarkers will be used for analysis.
  Short-term is defined as <= 26hours; biomarker kinetics are defined as >20% increase or decrease of a biomarker level at one point in time compared to the level at another point in time. The timestamp documented in the electronic health record will be used for analysis.
Short-term kinetics of bioimpedance | 4 days
  Outcome is the detection of kinetics of bioimpedance [Ohm] between at least two timestamps. The mean value within 1 h before the timestamp of the concomitant biochemical biomarkers will be used for analysis.
  Short-term is defined as <= 26hours; biomarker kinetics are defined as >20% increase or decrease of a biomarker level at one point in time compared to the level at another point in time. The timestamp documented in the electronic health record will be used for analysis.

SECONDARY OUTCOMES:
Correlation between C-reactive protein and body surface temperature | 4 days
  Outcome is the detection of a correlation between C-reactive protein [mg/L] and body surface temperature [°C].
  Correlations between physiological biomarkers and biochemical biomarkers will be analysed graphically and by Spearman's correlation coefficient.
Correlation between C-reactive protein and bioimpedance | 4 days
  Outcome is the detection of a correlation between C-reactive protein [mg/L] and bioimpedance [Ohm].
  Correlations between physiological biomarkers and biochemical biomarkers will be analysed graphically and by Spearman's correlation coefficient.
Correlation between procalcitonin and body surface temperature | 4 days
  Outcome is the detection of a correlation between procalcitonin [ng/mL] and body surface temperature [°C].
  Correlations between physiological biomarkers and biochemical biomarkers will be analysed graphically and by Spearman's correlation coefficient.
Correlation between procalcitonin and bioimpedance | 4 days
  Outcome is the detection of a correlation between procalcitonin [ng/mL] and bioimpedance [Ohm].
  Correlations between physiological biomarkers and biochemical biomarkers will be analysed graphically and by Spearman's correlation coefficient.
Correlation between interleukin-6 and body surface temperature | 4 days
  Outcome is the detection of a correlation between interleukin-6 [ng/L] and body surface temperature [°C].
  Correlations between physiological biomarkers and biochemical biomarkers will be analysed graphically and by Spearman's correlation coefficient.
Correlation between interleukin-6 and bioimpedance | 4 days
  Outcome is the detection of a correlation between interleukin-6 [ng/L] and bioimpedance [Ohm].
  Correlations between physiological biomarkers and biochemical biomarkers will be analysed graphically and by Spearman's correlation coefficient.
Correlation between ferritin and body surface temperature | 4 days
  Outcome is the detection of a correlation between ferritin [µg/L] and body surface temperature [°C].
  Correlations between physiological biomarkers and biochemical biomarkers will be analysed graphically and by Spearman's correlation coefficient.
Correlation between ferritin and bioimpedance | 4 days
  Outcome is the detection of a correlation between ferritin [µg/L] and bioimpedance [Ohm].
  Correlations between physiological biomarkers and biochemical biomarkers will be analysed graphically and by Spearman's correlation coefficient.
Correlation between NT-pro brain natriuretic peptide and body surface temperature | 4 days
  Outcome is the detection of a correlation between NT-pro brain natriuretic peptide [ng/L] and body surface temperature [°C].
  Correlations between physiological biomarkers and biochemical biomarkers will be analysed graphically and by Spearman's correlation coefficient.
Correlation between NT-pro brain natriuretic peptide and bioimpedance | 4 days
  Outcome is the detection of a correlation between NT-pro brain natriuretic peptide [ng/L] and bioimpedance [Ohm].
  Correlations between physiological biomarkers and biochemical biomarkers will be analysed graphically and by Spearman's correlation coefficient.
Correlation between high sensitive troponin T and body surface temperature | 4 days
  Outcome is the detection of a correlation high sensitive troponin T [ng/L] and body surface temperature [°C].
  Correlations between physiological biomarkers and biochemical biomarkers will be analysed graphically and by Spearman's correlation coefficient.
Correlation between high sensitive troponin T and bioimpedance | 4 days
  Outcome is the detection of a correlation high sensitive troponin T [ng/L] and bioimpedance [Ohm].
  Correlations between physiological biomarkers and biochemical biomarkers will be analysed graphically and by Spearman's correlation coefficient.
Correlation between lactate and body surface temperature | 4 days
  Outcome is the detection of a correlation between lactate [mg/dL] and body surface temperature [°C].
  Correlations between physiological biomarkers and biochemical biomarkers will be analysed graphically and by Spearman's correlation coefficient.
Correlation between lactate and bioimpedance | 4 days
  Outcome is the detection of a correlation between lactate [mg/dL] and bioimpedance [Ohm].
  Correlations between physiological biomarkers and biochemical biomarkers will be analysed graphically and by Spearman's correlation coefficient.
Correlation between blood pH and body surface temperature | 4 days
  Outcome is the detection of a correlation between blood pH and body surface temperature [°C].
  Correlations between physiological biomarkers and biochemical biomarkers will be analysed graphically and by Spearman's correlation coefficient.
Correlation between blood pH and bioimpedance | 4 days
  Outcome is the detection of a correlation between blood pH and bioimpedance [Ohm].
  Correlations between physiological biomarkers and biochemical biomarkers will be analysed graphically and by Spearman's correlation coefficient.